CLINICAL TRIAL: NCT03121092
Title: Should Ambulatory Surgery and Day of Surgery Admission Patients Discontinue Angiotensin Converting Enzyme Inhibitors (ACEI's) and Angiotension Receptor Blockers (ARB's) Preoperatively?
Brief Title: ACEI/ARB Study in Ambulatory and Day of Surgery Admission Patients
Acronym: ACE/ARB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulty with recruiting patients meeting the inclusion criteria the PI decided to retire this project.
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 303066-1
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Hypertension; Hypotension
MeSH Terms: conditions — Hypertension; Hypotension | interventions — Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Discontinue ACEI or ARB (No Intervention): Patients in this group will not take the ACE or ARB 24 hours prior to their procedure.
- Continue ACEI or ARB (Active Comparator): Patients in this group will take an ACE or ARB on the day of surgery.
  Interventions: Drug: ACEI or ARB

INTERVENTIONS:
Drug: ACEI or ARB — Angiotensin converting enzyme inhibitors (ACEI's) and Angiotensin receptor blockers (ARB's) - commonly used anti-hypertensive medications
  Arms: Continue ACEI or ARB

SUMMARY:
Angiotensin converting enzyme inhibitors (ACEI's) and Angiotensin receptor blockers (ARB's) are commonly used anti-hypertensive medications that may have implications on the management of a patient undergoing surgery. Limited research has looked at the effects of these medications on perioperative complications and mortality. Some studies conducted on small groups of inpatients with advanced vascular disease undergoing vascular surgery or coronary artery bypass grafting (CABG), suggest exacerbation of hypotension (low blood pressure) in patients who continued taking ACEI's or ARB's on the morning of their procedure. In addition, cases of low blood pressure (BP) that were refractory to standard treatment were reported. One recent retrospective study reported no difference in severe hypotension and only a modest difference in moderate hypotension managed by conventional treatment, but did not adequately address the risk of preoperative hypertension. A study recently published by the investigators (Twersky et al., 2014) in over 600 patients demonstrated no difference in preoperative hypertension in ambulatory surgery and same day admission patients. There has been limited data stratifying the degree of low BP based on severity but these were not done in ambulatory patients, and neither was the degree of high BP from discontinuing these medications addressed. As such, no uniform consensus has been reached and clinicians are unclear as to whether the reported inpatient findings are applicable to the outpatients, since they differ in many respects. The investigators propose to evaluate whether ACEI's and ARB's discontinued preoperatively have a negative impact on perioperative hemodynamics and patient outcome in a group of ambulatory and same day surgical patients. Similar to studies done on inpatients, the investigators will also evaluate patients receiving a standardized general anesthetic for hemodynamics following induction of anesthesia until surgical incision.

The investigators hypothesize that continuing ACEI's and ARB's in the preoperative period does not result in an increased risk of severe hypotension (low blood pressure) following induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 18
* patients scheduled to undergo any surgical procedure on an ambulatory basis or on a same day admission basis
* patients undergoing general anesthesia by Laryngeal Mask Airway (LMA)
* patients taking chronic ACEI or ARB drug treatment for hypertension for more than 6 weeks
* patients on diuretics and/or beta blockers and/or calcium channel blockers for hypertension in addition to the ACEI or ARB (alone or in combination) for hypertension may be included
* patients taking any cardiovascular medications may be included

Exclusion Criteria:

* patients taking both an ACEI and an ARB simultaneously
* patients taking ACEI or ARB for less than 6 weeks
* patients with uncontrolled hypertension during pre-surgical testing (PST) visit, defined as Systolic (SBP) > 180 or Diastolic (DBP) > 100 (Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure JNC 7)
* patients with history of unstable heart disease, refractory congestive heart failure, hypertensive stroke, mini stroke, stroke or heart attack within the past 6 months
* emergency surgery
* patients who are pregnant
* patients whose surgery requires endotracheal intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Presence of moderate hypotension | Through study completion, projected 2-3 years
  Presence of moderate hypotension (SBP<90 or a change of >30% from pre-induction baseline), in the intraoperative setting and in the post-anesthesia care unit
Presence of severe hypotension | Through study completion, projected 2-3 years
  Presence of severe hypotension (SBP<65) between induction and incision

SECONDARY OUTCOMES:
The prevalence of cancellation of surgery secondary to unstable BP | Through study completion, projected 2-3 years
The number and dose of medications to treat BP | Through study completion, projected 2-3 years
prevalence of adverse effects (increased length of stay in the PACU, unanticipated hospitalizations, myocardial ischemia, stroke, death) | Through study completion, projected 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ketan Shevde, MD, Principal Investigator — State University of New York - Downstate Medical Center; Rebecca Twersky, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Result] Twersky RS, Goel V, Narayan P, Weedon J. The risk of hypertension after preoperative discontinuation of angiotensin-converting enzyme inhibitors or angiotensin receptor antagonists in ambulatory and same-day admission patients. Anesth Analg. 2014 May;118(5):938-44. doi: 10.1213/ANE.0000000000000076. PMID 24681657